CLINICAL TRIAL: NCT06029829
Title: The Clinical Value of Peripheral Blood T Lymphocyte PD-1 Expression and T Cell Subset Distribution in the Immunotherapy of Advanced Primary HCC Patients.
Brief Title: The Clinical Significance of Peripheral Blood T Lymphocyte PD-1 Expression and T Cell Subset Distribution.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xin-Hua Xu (Other)
Responsible Party: Sponsor-Investigator, Xin-Hua Xu, professor, China Three Gorges University, Yichang, China
Organization: China Three Gorges University, Yichang, China (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTGU008
Record Dates: First submitted 2023-08-26; First posted 2023-09-08 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Immunomonotherapy plus Chemotherapy plus Anti-angiogenesis Therapy (Experimental): Any first-line treatment that includes immunotherapy、 Chemotherapy and Anti-angiogenesis Therapy
  Interventions: Drug: Sintilimab

INTERVENTIONS:
Drug: Sintilimab — Any first-line treatment that includes immunotherapy、 Chemotherapy and Anti-angiogenesis Therapy

SUMMARY:
Providing more theoretical basis for the prediction of the efficacy of advanced HCC and helping select better advantaged population of HCC immunotherapy to maximize the benefits of patients By exploring the relationship between the changes of PD-1 expression in peripheral blood T lymphocytes and the clinical efficacy before and after the use of PD-1 / PD-L1 inhibitors.

DETAILED DESCRIPTION:
Exploring the expression of peripheral blood T lymphocyte PD-1 from an immunological perspective as a potential reference marker for selecting immunotherapy in advanced HCC patients, and elucidating the relationship between the level of peripheral blood T lymphocyte PD-1 expression and survival outcomes after receiving immunotherapy. Additionally, investigating whether there is consistency between the expression levels of PD-1 and PD-L1 and their impact on patients. Furthermore, exploring the correlation between the distribution of T cell subsets and the efficacy of immunotherapy to provide new theoretical evidence for the selection of target populations for immunotherapy and new clinical screening indicators for patient prognosis assessment.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate in the clinical study, fully understand and be informed about the study, and sign the informed consent form;
* Age between 18 and 75 years, male or female;
* Strictly meet the clinical diagnostic criteria for hepatocellular carcinoma (HCC), confirmed by histology or cytology, with at least one lesion meeting the RECIST 1.1 criteria on CT or MRI examination;
* No prior targeted therapy, immunotherapy, or systemic chemotherapy for liver cancer before admission;
* Child-Pugh A liver function; Barcelona Clinic Liver Cancer (BCLC) stage B or C;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1;
* Normal function of major organs;
* Expected survival time of at least 12 weeks or more.

Exclusion Criteria:

* Patients who have not previously received treatment with Sintilimab or any other PD-L1 or PD-1 antagonist;
* Patients with any active autoimmune disease or a history of autoimmune disease, or a history of immunodeficiency;
* Patients requiring the use of immunosuppressive drugs;
* Known history of allergy to the formulation of Sintilimab or any other component of the antibody formulation;
* Patients with other malignant tumors.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-12 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Compare Progression Free Survival (PFS) Regimen using RECIST 1.1. | 24 months
  PFS was defined as the time between the date of randomization and the date of first documented disease progression or death, whichever occurs first. Disease progression was determined based on investigator assessment using response evaluation criteria In solid tumors (RECIST) v1.1.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medical Oncology, Central Hospital of Yichang City, the First Clinical Medical College of Three Gorges University, Yichang, Hubei, China